CLINICAL TRIAL: NCT03930082
Title: Application of Frailty Assessment in Elderly Patients Undergoing Gastrointestinal Surgery
Brief Title: Frailty Assessment of Patients With Gastrointestinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ziqiang Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Ziqiang Wang,MD, Clinical professor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: FA-PGS-2019
Record Dates: First submitted 2019-04-04; First posted 2019-04-29 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Gastrointestinal Disease; Frail Elderly Syndrome
Keywords: Gastrointestinal surgery; Frailty; Elder patient; Complication
MeSH Terms: conditions — Gastrointestinal Diseases; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Frailty Index Scale — We will evaluate the frailty with a Frailty Index Scale in elderly patients undergoing gastrointestinal surgery.

SUMMARY:
Patients aged 65 or older under gastrointestinal surgery will be enrolled，the investigators will assess the frailty of these patients by Frailty Index Scale and explore the correlation between the frailty and perioperative adverse events.

DETAILED DESCRIPTION:
Patients will be assessed by specially trained doctors or nurses after admission, including daily living ability, physiological function, social-psychological status, comorbidities, mental state, grip strength, walking speed. After the assessment, the patients' frailty index was obtained. Moreover, the operation time, intraoperative bleeding loss, perioperative complications, length of stay, hospitalization expenses, readmission rate within 30 days, mortality within 30 days and other outcome indicators of these patients will be recorded.

The Main purposes of present study are to verify the feasibility of applying Frailty Index (FI) to assess the degree of frailty in elderly patients undergoing gastrointestinal surgery, compare the difference of perioperative adverse events in elderly patients with different degrees of frailty，find potential indicators for evaluating and predicting the safety of surgery in elderly patients, and provide reference data for the determination of future assessment tools of frailty.

The secondary objective is to compare the quality of life and long-term prognosis(only for patients with cancers,including recurrence free survival and overall survival) of elderly patients with different degrees of frailty after gastrointestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age not less than 65 years;
* undergoing operation in gastrointestinal surgery of West China hospital due to gastrointestinal disease.

Exclusion Criteria:

* Those who did not undergo surgery for various reasons;
* Death before operation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged 65 years or older who undergo gastrointestinal surgery in West China Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
operative time | 2 year
  From the beginning of the skin incision to the end of the last incision was From the beginning of the skin incision to the end of the suture of last incision
Blood loss | 2 year
  intraoperative blood loss
Intraoperative complications | 2 year
  Including all the complications in the procedure
postoperative complications | 2 year
  including incision infection，anastomotic leakage，respiratory infection, postoperative bleeding and so on.
The length of stay in intensive care unit (ICU) | 2 year
  Time form entry to ICU to return to general ward after the condition is stable.
The length of hospitalization | 2 year
  Time from admission to discharge
Hospital costs | 2 year
  Cost of diagnosis and treatment during hospitalization
Readmission rate within 30 days | 2 year
  The proportion of patients who are re-hospitalized for postoperative complications after 30 days of discharge in all subjects.
Mortality within 30 days | 2 year
  death rate within 30 days after surgery in all patients after operation

SECONDARY OUTCOMES:
Recurrence-free Survival (RFS) | 2 year
  RFS is the abbreviation of recurrence-free survival, which refers to the duration from postoperation to tumor recurrence (Only for patients with cancers).
Overall survival (OS) | 2 year
  OS is the abbreviation of overall survival , which refers to the duration from postoperation to death of the subjects (Only for patients with cancers).

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, MD,PHD, Study Chair — Department of Gastrointestinal Surgery, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No